CLINICAL TRIAL: NCT07057726
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial Evaluating the Safety, Tolerability, and Pharmacokinetics of SSS39 Injection by Single Intravenous Infusion in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SSS39 Injection in Healthy Chinese Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: SYSS-SSS39-UND-I-01
Record Dates: First submitted 2025-02-06; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Safety and Tolerability in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Low-dose Group
  Interventions: Drug: SSS39
- group 2 (Experimental): high dose Group
  Interventions: Drug: SSS39

INTERVENTIONS:
Drug: SSS39 — Single oral administration of SSS39
  Arms: group 1
Drug: SSS39 — Single oral administration of SSS39
  Arms: group 2

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetics of SSS39 injection in healthy Chinese subjects

DETAILED DESCRIPTION:
This study was a single-administration, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK profile, immunogenicity, and effects on Treg cells and cytokines of SSS39 injection in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy subjects aged 18-45 years old (including boundary values), regardless of gender;
* 2. Subjects voluntarily participate in clinical trials and sign informed consent;
* 3. Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) between 19-28 kg/m2 (including the cut-off value);

Exclusion Criteria:

* 1.Have a clear history of drug or food allergy, or are known to have an allergic reaction to Sirolimus, polyethylene glycol and any excipients of this product, including lactose intolerance;
* 2.Subjects who have received any other drug that acts on the mammalian target protein of rapamycin (mTOR);
* 3. within 14 days prior to administration of the investigational product (or five half-lives of CYP3A4/P-gp inhibitors/inducers, whichever is longer), or anticipated use of a known major CYP3A4/P-gp inhibitor or major CYP3A4/P-gp inducer (including natural products) during the trial, Such as St. John's wort or grapefruit juice);
* 4.Abnormal results of sedimentation, abdominal B-ultrasonography, kidney B-ultrasonography or superficial lymph node B-ultrasonography during the screening period were judged by researchers to be clinically significant;
* 5. Acute or chronic systemic infection or local infection within 2 weeks before screening;
* 6. Previous or current history of autoimmune disease, immune deficiency, or history of organ transplantation, or/and use of immunomodulatory or immunosuppressive drugs within 6 months prior to screening;
* 7. Those who have had major surgery or have not fully recovered from any previous invasive procedure within 4 weeks prior to dosing;
* 8. Have syphilis (positive for treponema pallidum antibodies) or AIDS (positive for HIV antibodies), or active hepatitis C (positive for hepatitis C virus antibodies and positive for hepatitis C virus [HCV]RNA results), or active hepatitis B (positive for hepatitis B surface antigen and hepatitis B virus [HBV] DNA above the lower limit of quantitative values);
* 9. Patients with past or present history of any clinically serious diseases, including but not limited to digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, neuropsychiatric system, blood system, etc. (except those considered by researchers to be eligible for inclusion);
* 10. Past or present history of malignant tumors;
* 11. Use of any drug (including prescription, over-the-counter, Chinese herbal, etc.) or supplement within 2 weeks prior to administration (if determined by the investigator, the time interval between the drug used and the beginning of administration of this trial > 5 half-lives, corresponding subjects can also be enrolled);
* 12. Those who received live vaccines within 1 month before administration or planned to receive live vaccines during the study period, including but not limited to: measles, mumps, rubella, chickenpox, yellow fever, rabies, BCG, typhoid vaccine, etc.;
* 13.Previous alcohol abuse or regular alcohol consumption in the 6 months prior to the test (drinking more than 14 units of alcohol per week, 1 unit =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine) or a positive alcohol breath test (breath alcohol content > 0.0 mg/100 mL), or those who cannot abstain from alcohol during the trial;
* 14.Those who test positive for one or more drug addiction and drug abuse tests, or have a history of drug abuse/dependence or drug abuse within the previous year;
* 15. habitual excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups a day, 1 cup =200 mL), and/or ingestion of any food or beverage containing caffeine, alcohol, xanthine and other ingredients (such as coffee, strong tea, chocolate, etc.) within 48 hours before administration;
* 16.Smokers who smoked more than 5 cigarettes per day in the 3 months before screening and those who could not smoke during the whole test period;
* 17. Participants who have participated in any drug clinical trial and taken experimental drugs, or participated in device clinical trial and used experimental devices within 3 months before screening;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerance of SSSS55 | Day 50
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- SSS39, Beijing, China

IPD SHARING:
Plan to Share IPD: No